CLINICAL TRIAL: NCT04539730
Title: Does the Addition of Liposomal Bupivacaine to the Adductor Canal Block Impact Narcotic Use After Primary Total Knee Arthroplasty: a Prospective, Blind Randomized Control Trial
Brief Title: Liposomal Bupivacaine in Adductor Canal Blocks (ACB)
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Did not acquire funding to pursue study
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Jaime Carvajal Alba, Assistant Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20200003
Record Dates: First submitted 2020-08-31; First posted 2020-09-07 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Arthroplasty Complications; Adductor Canal Block; Peripheral Nerve Block; Opioid Use
Keywords: Total knee arthroplasty

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and study team members involved in data collection and data processing will be blinded to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ropivacaine Standard of Care Group (Active Comparator): Participants undergoing elective Total Knee Arthoplasty (TKA) surgery that are randomized to the control group will undergo an ultrasound-guided Adductor Canal Block (ACB) with standard of care (SoC) Ropivacaine post TKA surgery.
  Interventions: Procedure: Drug: SoC Ropivacaine
- Liposomal Bupivacaine Intervention Group (Experimental): Participants undergoing elective TKA surgery that are randomized to the intervention group will undergo an ultrasound-guided ACB with Liposomal Bupivacaine post TKA surgery.
  Interventions: Drug: Liposomal bupivacaine; Procedure: Drug: SoC Ropivacaine

INTERVENTIONS:
Drug: Liposomal bupivacaine — 266 mg or 20 ml Liposomal Bupivacaine injectable solution
  Other Names: Exparel
  Arms: Liposomal Bupivacaine Intervention Group
Procedure: Drug: SoC Ropivacaine — 0.5% (5mg/mL) 20 mL single dose SOC anesthetic Ropivacaine.

SUMMARY:
The purpose of this study is to evaluate whether liposomal bupivacaine is superior to normal bupivacaine in terms of providing better pain control postoperatively after total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is scheduled for elective unilateral primary TKA
2. The subject is ≥ 18 years
3. The subject's primary anesthesia care team has planned for a neuraxial anesthetic (i.e. spinal, epidural or combined-spinal epidural)
4. The patient consents for an adductor canal block
5. Willing and able to sign an informed consent.

Exclusion Criteria:

1. Patients unwilling or unable to consent to participate in the study.
2. Prisoners.
3. Pregnancy.
4. Reported to have mental illness or belonging to a vulnerable population.
5. Subject is < 18 years of age.
6. Patients receiving general anesthesia for the total knee arthroplasty.
7. Subject has impaired decision-making capacity per discretion of the Investigator.
8. Any condition for which the primary anesthesia care team deems neuraxial anesthesia inappropriate.
9. Significant pre-existing neuropathy on the operative limb.
10. Significant chronic pain disorders (i.e. fibromyalgia, complex regional pain syndrome I & II, among others).
11. Subject has sustained a significant trauma to the operative knee.
12. Chronic Opioid Use (daily or almost daily use of opioids for > 3 months).
13. Known hypersensitivity and/or allergies to local anesthetics.
14. Previous surgery on the affected knee excluding arthroscopic or open meniscectomy.
15. Patients with impaired renal function such that they cannot receive IV Toradol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Opioid Use | Up to 2 weeks
  Opioid use after SoC TKA surgery will be evaluated as morphine milligram equivalents

SECONDARY OUTCOMES:
Distance Ambulated with physical therapist | Up to 5 days
  Average daily distance ambulated using the 6 minute walk test
Length of hospitalization | Up to 5 days
  Number of days of hospitalization after elective admission for TKA surgery
Incidence of events of PONV | Up to 5 days
  Incidence of post-operative nausea and vomiting (PONV) will be reported throughout the duration of hospitalization
Number of participants requiring narcotic prescriptions | 2 weeks
  The number of participants that require further narcotic prescriptions will be reported
Incidence of urinary retention from narcotic use | 2 Weeks
  Incidence of urinary retention from narcotic use will be measured via the need for urethral catheterization.
Post-Operative Pain Score | Up to 5 days
  Post-Operative Pain will be measured via a self-reported Visual Analog Scale (VAS) score. The VAS Pain score ranges from 1-10 with 1 being free of pain and 10 being the most pain.
Patient Satisfaction as per the Knee Society Score | Up to Week 6
  The Knee society score has a total score ranging from 100-0. Scores between 100 and 85 points are considered excellent results, scores between 84 and 70 points are considered good results. Scores between 69 and 60 points are considered fair, and scores less than 60 are considered poor results

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Carvajal, MD, Principal Investigator — University of Miami

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grevstad U, Mathiesen O, Valentiner LS, Jaeger P, Hilsted KL, Dahl JB. Effect of adductor canal block versus femoral nerve block on quadriceps strength, mobilization, and pain after total knee arthroplasty: a randomized, blinded study. Reg Anesth Pain Med. 2015 Jan-Feb;40(1):3-10. doi: 10.1097/AAP.0000000000000169. PMID 25376972
- [Background] Thacher RR, Hickernell TR, Grosso MJ, Shah R, Cooper HJ, Maniker R, Brown AR, Geller J. Decreased risk of knee buckling with adductor canal block versus femoral nerve block in total knee arthroplasty: a retrospective cohort study. Arthroplast Today. 2017 Apr 15;3(4):281-285. doi: 10.1016/j.artd.2017.02.008. eCollection 2017 Dec. PMID 29204497
- [Background] Singh PM, Borle A, Trikha A, Michos L, Sinha A, Goudra B. Role of Periarticular Liposomal Bupivacaine Infiltration in Patients Undergoing Total Knee Arthroplasty-A Meta-analysis of Comparative Trials. J Arthroplasty. 2017 Feb;32(2):675-688.e1. doi: 10.1016/j.arth.2016.09.042. Epub 2016 Oct 8. PMID 28029532
- [Background] Schroer WC, Diesfeld PG, LeMarr AR, Morton DJ, Reedy ME. Does Extended-Release Liposomal Bupivacaine Better Control Pain Than Bupivacaine After Total Knee Arthroplasty (TKA)? A Prospective, Randomized Clinical Trial. J Arthroplasty. 2015 Sep;30(9 Suppl):64-7. doi: 10.1016/j.arth.2015.01.059. Epub 2015 Jun 3. PMID 26117072
- [Background] Jain RK, Porat MD, Klingenstein GG, Reid JJ, Post RE, Schoifet SD. The AAHKS Clinical Research Award: Liposomal Bupivacaine and Periarticular Injection Are Not Superior to Single-Shot Intra-articular Injection for Pain Control in Total Knee Arthroplasty. J Arthroplasty. 2016 Sep;31(9 Suppl):22-5. doi: 10.1016/j.arth.2016.03.036. Epub 2016 Mar 26. PMID 27113945
- [Background] Bagsby DT, Ireland PH, Meneghini RM. Liposomal bupivacaine versus traditional periarticular injection for pain control after total knee arthroplasty. J Arthroplasty. 2014 Aug;29(8):1687-90. doi: 10.1016/j.arth.2014.03.034. Epub 2014 Apr 4. PMID 24793570
- [Background] Haas E, Onel E, Miller H, Ragupathi M, White PF. A double-blind, randomized, active-controlled study for post-hemorrhoidectomy pain management with liposome bupivacaine, a novel local analgesic formulation. Am Surg. 2012 May;78(5):574-81. doi: 10.1177/000313481207800540. PMID 22546131
- [Background] Surdam JW, Licini DJ, Baynes NT, Arce BR. The use of exparel (liposomal bupivacaine) to manage postoperative pain in unilateral total knee arthroplasty patients. J Arthroplasty. 2015 Feb;30(2):325-9. doi: 10.1016/j.arth.2014.09.004. Epub 2014 Sep 16. PMID 25282071
- [Background] Zhao B, Ma X, Zhang J, Ma J, Cao Q. The efficacy of local liposomal bupivacaine infiltration on pain and recovery after Total Joint Arthroplasty: A systematic review and meta-analysis of randomized controlled trials. Medicine (Baltimore). 2019 Jan;98(3):e14092. doi: 10.1097/MD.0000000000014092. PMID 30653126
- See also: Related Info — http://www.exparel.com